CLINICAL TRIAL: NCT02171494
Title: Bioequivalence of 2x5 mg of IVAX Warfarin /Formulation Tablet Compared to 10 mg of Coumadin /Formulation Tablet Following Oral Administration in Healthy Male Volunteers (an Open-label, Randomised, Single-dose, Two-treatment, Two-sequence Crossover Study) Under Fasted Conditions
Brief Title: Bioequivalence of IVAX Warfarin Tablets and Coumadin Brand Warfarin Tablets in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.68
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy

ARMS (2):
- IVAX warfarin (Experimental): Treatment A: IVAX warfarin
  Interventions: Drug: IVAX Warfarin
- BMS coumadin (Active Comparator): Treatment B: BMS coumadin tablets
  Interventions: Drug: BMS Coumadin

INTERVENTIONS:
Drug: IVAX Warfarin
  Arms: IVAX warfarin
Drug: BMS Coumadin
  Arms: BMS coumadin

SUMMARY:
To establish the bioequivalence of 2x5 mg of IVAX warfarin /formulation tablet vs. 10 mg of Coumadin / formulation tablet

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (blood pressure, pulse rate, temp), 12-lead electrocardiogram, clinical laboratory tests, without clinically significant abnormal findings
* Age ≥ 18 and Age ≤ 45 years
* Body Mass Index (BMI) ≥ 18.0 and BMI ≤ 30.0 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and the local legislation

Exclusion Criteria:

* A history of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the investigator, would jeopardize the safety of the subject or impact the validity of the study results
* A history of allergic or adverse responses to warfarin or any comparable or similar product
* Subjects who (for whatever reason) had been on an abnormal diet or had substantial changes in eating habits within 30 days prior to study initiation
* Subjects could not have made a blood donation of one pint or more within 30 days prior to study initiation
* Subjects could not have made a plasma donation within 14 days of study initiation
* Participation in a clinical trial within 30 days prior to study initiation
* Use of any over-the-counter (OTC) medication, including vitamins, herbal products, and dietary supplements, within 7 days prior to or during the study
* Use of any prescription medication within 7 days prior to or during the study
* Treatment with any known enzyme altering drugs such as barbiturates, phenothiazines, cimetidine, carbamazepine, phenytoin, rifampin, rifabutin, glucocorticoids, diltiazem, ketoconazole, MAOI (monoamine oxidase inhibitor), antidepressants, neuroleptics, verapamil, quinidine, erythromycin, etc., within 30 days prior to or during the study
* Smoking or use of tobacco products within 6 months prior to or during the study. Smoking status was verified by a urine cotinine screen.
* Female subjects
* Positive blood screen for Human Immunodeficiency Virus, Hepatitis B, or Hepatitis C
* Positive screen for alcohol, drugs of abuse, or cotinine and history or presence of alcoholism or drug abuse within 6 months prior to the study start
* Subjects could not have taken aspirin or any aspirin-containing medications or any antiplatelet or anticoagulant medication within 7 days prior to the study, for the duration of the study and for 14 days after the last dose of study medication
* aPTT (activated partial thromboplastin time) or INR (international normalized ratio) results unacceptable to principal investigator
* Inability to comply with dietary regimen of trial site

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
AUC0-infinity (area under the concentration-time curve over the time interval from 0 extrapolated to infinity) | pre-dose and 0:15, 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30, 4:00, 5:00, 6:00, 8:00,10:00 12:00, 24:00, 36:00, 48:00, 72:00, 96:00, 120:00, 144:00, 168:00, 192:00 and 216:00 hours after dosing on day 1 and day 22
Cmax (maximum measured concentration of the analyte in plasma) | pre-dose and 0:15, 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30, 4:00, 5:00, 6:00, 8:00,10:00 12:00, 24:00, 36:00, 48:00, 72:00, 96:00, 120:00, 144:00, 168:00, 192:00 and 216:00 hours after dosing on day 1 and day 22

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve over the time interval from 0 to the time of the last quantifiable data point) | pre-dose and 0:15, 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30, 4:00, 5:00, 6:00, 8:00,10:00 12:00, 24:00, 36:00, 48:00, 72:00, 96:00, 120:00, 144:00, 168:00, 192:00 and 216:00 hours after dosing on day 1 and day 22
tmax (time from dosing to the maximum concentration) | pre-dose and 0:15, 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30, 4:00, 5:00, 6:00, 8:00,10:00 12:00, 24:00, 36:00, 48:00, 72:00, 96:00, 120:00, 144:00, 168:00, 192:00 and 216:00 hours after dosing on day 1 and day 22
λz (terminal rate constant in plasma) | pre-dose and 0:15, 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30, 4:00, 5:00, 6:00, 8:00,10:00 12:00, 24:00, 36:00, 48:00, 72:00, 96:00, 120:00, 144:00, 168:00, 192:00 and 216:00 hours after dosing on day 1 and day 22
t1/2 (terminal half-life of the analyte in plasma) | pre-dose and 0:15, 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30, 4:00, 5:00, 6:00, 8:00,10:00 12:00, 24:00, 36:00, 48:00, 72:00, 96:00, 120:00, 144:00, 168:00, 192:00 and 216:00 hours after dosing on day 1 and day 22
MRTpo (mean residence time of the analyte in the body after oral administration) | pre-dose and 0:15, 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30, 4:00, 5:00, 6:00, 8:00,10:00 12:00, 24:00, 36:00, 48:00, 72:00, 96:00, 120:00, 144:00, 168:00, 192:00 and 216:00 hours after dosing on day 1 and day 22
CL/F (apparent clearance after extravascular administration) | pre-dose and 0:15, 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30, 4:00, 5:00, 6:00, 8:00,10:00 12:00, 24:00, 36:00, 48:00, 72:00, 96:00, 120:00, 144:00, 168:00, 192:00 and 216:00 hours after dosing on day 1 and day 22
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | pre-dose and 0:15, 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 3:30, 4:00, 5:00, 6:00, 8:00,10:00 12:00, 24:00, 36:00, 48:00, 72:00, 96:00, 120:00, 144:00, 168:00, 192:00 and 216:00 hours after dosing on day 1 and day 22